CLINICAL TRIAL: NCT05065086
Title: Single Modality Trans Oral Robotic Surgery for Primary Oropharyngeal Cancer: Exploring the Impact of Surgical Margins on Local Disease Recurrence
Acronym: STORM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5370
Record Dates: First submitted 2021-09-06; First posted 2021-10-01 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Primary OPSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective observational cohort study investigating Single modality Trans Oral Robotic surgery for primary oropharyngeal cancer: exploring the impact of surgical Margins on local disease recurrence.

DETAILED DESCRIPTION:
The STORM study will examine transoral surgery performed before 31st July 2019. STORM is a retrospective observational cohort study, involving international centres performing TORS for primary OPSCC.

The main aim of this study is to explore the impact of surgical margins on local disease recurrence in primary oropharyngeal squamous cell carci-noma treated with transoral robotic surgery (TORS) without adjuvant therapy.

The primary objective is to report local recurrence-free survival. The primary endpoint will be Local recurrence-free survival time.

The secondary objectives are to report overall survival, disease-specific survival and disease-free survival, and to report post-operative haemor-rhage rates. The secondary endpoints include Overall survival time, Dis-ease-specific survival time, Disease-free survival time, Post-operative haemorrhage time.

Exploratory objective to identify a clinically relevant cut-off for surgical margins as a predictor of local disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Primary OPSCC.
* Index cancer treated with TORS without adjuvant therapy.
* Any post-operative TNM classification.
* TORS performed on or before 31st July 2019.

Exclusion Criteria:

* TORS preformed for diagnostic or palliative intentions.
* Known distant metastasis at time of TORS.
* Nasopharyngeal and thyroid cancers.
* Patients undergoing neoadjuvant or adjuvant chemotherapy, biotherapy, immunotherapy or radiotherapy to either the neck or primary site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Primary OPSCC with Index cancer treated with TORS, without adjuvant therapy, on or before 31st July 2019.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Local recurrence-free survival time | At 2 years

SECONDARY OUTCOMES:
Overall survival time | At 2 and 5 years
Disease-specific survival time | At 2 and 5 years
Disease-free survival time | At 2 and 5 years
Post-operative haemorrhage time | Within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No